CLINICAL TRIAL: NCT00547586
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, Parallel-Group Study of Oral MOA-728 for the Treatment of Opioid- Induced Bowel Dysfunction in Subjects With Chronic Nonmalignant Pain
Brief Title: Study Evaluating Oral MOA-728 For The Treatment Of OIBD In Subjects With Chronic Non-Malignant Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3200A3-2201
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Other: placebo
- 150 mg (Experimental)
  Interventions: Drug: N-methylnaltrexone bromide (MOA-728)
- 300 mg (Experimental)
  Interventions: Drug: N-methylnaltrexone bromide (MOA-728)
- 450 mg (Experimental)
  Interventions: Drug: N-methylnaltrexone bromide (MOA-728)
- 600 mg (Experimental)
  Interventions: Drug: N-methylnaltrexone bromide (MOA-728)

INTERVENTIONS:
Drug: N-methylnaltrexone bromide (MOA-728) — Oral
  Arms: 150 mg; 300 mg; 450 mg; 600 mg
Other: placebo — placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and dose-response relationship of N-methylnaltrexone bromide (MOA-728) by observing spontaneous bowel movements in subjects with chronic pain, which is not due to malignant cancer, and who have opioid-induced bowel dysfunction (OIBD).

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients with opioid-induced bowel dysfunction and chronic pain, which is not due to malignant cancer.
* Taking oral, transdermal, intravenous, or subcutaneous opioids.
* Willingness to discontinue all pre-study laxative therapy and use only study permitted rescue laxatives.

Exclusion Criteria:

* History of chronic constipation before the initiation of opioid therapy.
* Other GI disorders known to affect bowel transit.
* Women who are pregnant, breast-feeding, or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (39):
- United States (39):
  - Mobile, Alabama
  - Litchfield Park, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Garden Grove, California
  - Long Beach, California
  - Los Angeles, California
  - Murrieta, California
  - San Diego, California
  - Chiefland, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Largo, Florida
  - Naples, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - Spring Hill, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Sunset, Louisiana
  - Elkridge, Maryland
  - Brockton, Massachusetts
  - Cadillac, Michigan
  - Traverse City, Michigan
  - Biloxi, Mississippi
  - Ocean Springs, Mississippi
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Dayton, Ohio
  - Toledo, Ohio
  - Medford, Oregon
  - Chattanooga, Tennessee
  - Beaumont, Texas
  - Colleyville, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Alexandria, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 150 mg | 300 mg | 450 mg | 600 mg
Started | 33 | 7 | 14 | 33 | 35
Completed | 28 | 6 | 13 | 27 | 32
Not Completed | 5 | 1 | 1 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 150 mg | 300 mg | 450 mg | 600 mg | Total
Number analyzed (Participants) | 33 | 7 | 14 | 33 | 35 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (8.75) | 48.43 (6.80) | 52.43 (8.56) | 51.21 (12.24) | 49.51 (11.25) | 49.84 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 5 | 5 | 24 | 18 | 74
  Male | 11 | 2 | 9 | 9 | 17 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Spontaneous Bowel Movement (SBM) Within 1, 2, 3, 4, and 6 Hours of Treatment
Time Frame: 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 150 mg | 300 mg | 450 mg | 600 mg
Number analyzed (Participants) | 33 | 7 | 14 | 33 | 35
Participants
  Within 1 hour of 1st dose | 0 | 0 | 0 | 7 | 2
  Within 2 hours of 1st dose | 1 | 1 | 1 | 9 | 5
  Within 3 hours of 1st dose | 3 | 1 | 2 | 13 | 9
  Within 4 hours of 1st dose | 3 | 1 | 4 | 15 | 14
  Within 6 hours of 1st dose | 6 | 1 | 4 | 15 | 17

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Placebo | 150 mg | 300 mg | 450 mg | 600 mg
All-Cause Mortality (participants affected / at risk) | 15/33 | 3/7 | 4/14 | 13/33 | 18/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/7 | 0/14 | 1/33 | 3/35
Other Adverse Events (participants affected / at risk) | 10/33 | 3/7 | 4/14 | 9/33 | 6/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | 150 mg (N=7) | 300 mg (N=14) | 450 mg (N=33) | 600 mg (N=35)
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lymphedema (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Cellulitis staphyloccocal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | 150 mg (N=7) | 300 mg (N=14) | 450 mg (N=33) | 600 mg (N=35)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distention (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2
Flatulence (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.